CLINICAL TRIAL: NCT04241575
Title: Identification of Fatty Liver With Advanced Fibrosis in Patients With Type 2 Diabetes Using Simple Fibrosis Scores and Electronic Reminder Messages: A Randomized Controlled Trial
Brief Title: Identification of Fatty Liver With Advanced Fibrosis in Type 2 Diabetes Using Simple Fibrosis Scores and Electronic Reminder Messages
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Vincent WS Wong, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Screening
Other Study IDs: NAFLD-NIT-RCT
Record Dates: First submitted 2020-01-23; First posted 2020-01-27 (Actual); Results first posted 2024-08-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Fatty Liver, Nonalcoholic; Diabetes Mellitus, Type 2
Keywords: Fatty liver; Non-invasive assessment; Case identification
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Diabetes Mellitus, Type 2; Fatty Liver

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): For patients in the intervention group, we will calculate the fibrosis scores. For patients with increased fibrosis scores, we will type the following pop-up message in our electronic clinical management system:
  "This patient has high Fibrosis-4 index (and/or AST-to-platelet ratio index) of xxx suggestive of significant liver fibrosis. Please consider referring the patient to the hepatology clinic or arranging further test such as FibroScan."
  The reminder message will pop up when physicians see the patient at the clinic and use the electronic clinical management system. The message will remain active for one year. Although the message is entered manually at this stage, the arrangement mimics an automated computer system. If the study results are positive, the next step is to modify the system to automate the process.
  Interventions: Diagnostic Test: Simple fibrosis scores and electronic reminder messages
- Control group (No Intervention): Patients in the control group will undergo the same assessments as patients in the intervention group. Although physicians will have access to the raw liver biochemistry results and platelet count, the fibrosis score results will not be specifically shown, and there will be no electronic reminder messages regardless of the fibrosis scores. This is to mimic usual care when there is no dedicated care model for case identification.

INTERVENTIONS:
Diagnostic Test: Simple fibrosis scores and electronic reminder messages — For patients in the intervention group, we will calculate the fibrosis scores. For patients with increased fibrosis scores, we will type the following pop-up message in our electronic clinical management system:
  "This patient has high Fibrosis-4 index (and/or AST-to-platelet ratio index) of xxx suggestive of significant liver fibrosis. Please consider referring the patient to the hepatology clinic or arranging further test such as FibroScan."
  The reminder message will pop up when physicians see the patient at the clinic and use the electronic clinical management system. The message will remain active for one year. Although the message is entered manually at this stage, the arrangement mimics an automated computer system. If the study results are positive, the next step is to modify the system to automate the process.
  Arms: Intervention group

SUMMARY:
Nonalcoholic fatty liver disease (NAFLD) is currently the most common chronic liver disease worldwide and is a major cause of cirrhosis and liver cancer in Western countries. Because of its close association with obesity and diabetes, most patients are seen by primary care physicians and endocrinologists rather than hepatologists. Previous studies have shown that NAFLD is under-recognized outside specialist settings. As a result, many patients are undiagnosed and not receiving specific treatments. With this background, we aim to test the hypothesis that the use of simple fibrosis scores as part of a diabetes complications screening program followed by electronic reminder messages is more effective than usual care in prompting physicians to correctly identify patients with suspected NAFLD and advanced liver fibrosis for specialist referral or further liver assessment. Our secondary aim is to test the hypothesis that the use of fibrosis scores and electronic reminder messages can increase the number of patients with confirmed diagnosis of advanced liver fibrosis.

DETAILED DESCRIPTION:
This will be a parallel group, randomized controlled trial. Patients fulfilling the inclusion and exclusion criteria above will be randomized 1:1 to two groups. Randomization will be carried out through the use of computer-generated list of random numbers in variable blocks of 4 to 10. Concealment of group allocation will be achieved through putting the group allocation cards in consecutively-numbered and sealed envelopes. The patients and physicians will know that the patients are in the intervention group if they see the reminder messages. When they do not see a reminder message, there will not be a specific indicator of whether the patient is in the control group or in the intervention group but having low fibrosis scores. Furthermore, the outcome assessors will be blinded to the group assignment.

For patients in the intervention group, we will calculate the fibrosis scores. For patients with increased fibrosis scores, we will type the following pop-up message in our electronic clinical management system:

"This patient has high Fibrosis-4 index (and/or AST-to-platelet ratio index) of xxx suggestive of significant liver fibrosis. Please consider referring the patient to the hepatology clinic or arranging further test such as FibroScan."

The reminder message will pop up when physicians see the patient at the clinic and use the electronic clinical management system. The message will remain active for one year. Although the message is entered manually at this stage, the arrangement mimics an automated computer system. If the study results are positive, the next step is to modify the system to automate the process.

Patients in the control group will undergo the same assessments as patients in the intervention group. Although physicians will have access to the raw liver biochemistry results and platelet count, the fibrosis score results will not be specifically shown, and there will be no electronic reminder messages regardless of the fibrosis scores. This is to mimic usual care when there is no dedicated care model for case identification.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-70 years
* Having type 2 diabetes
* Provided informed written consent

Exclusion Criteria:

* Type 1 diabetes
* Already receiving specialist care by gastroenterologists or hepatologists
* Current or past history of hepatocellular carcinoma or liver decompensation
* Active malignancies other than hepatocellular carcinoma, unless in complete remission for more than 5 years

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1061 (Actual)
Dates: Start 2020-05-19 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2023-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Wong, MD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
Selected data may be shared with other researchers upon reasonable request.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 1-5 years after the publication of the full paper.
Access Criteria: Researchers with clear plans of collaboration and analysis

REFERENCES:
- [Derived] Zhang X, Yip TC, Wong GL, Leow WX, Liang LY, Lim LL, Li G, Ibrahim L, Lin H, Lai JCT, Chim AM, Chan HLY, Kong AP, Chan WK, Wong VW. Clinical care pathway to detect advanced liver disease in patients with type 2 diabetes through automated fibrosis score calculation and electronic reminder messages: a randomised controlled trial. Gut. 2023 Nov 24;72(12):2364-2371. doi: 10.1136/gutjnl-2023-330269. PMID 37549979

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention Group | Control Group
Started | 533 | 528
Completed | 533 | 528
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Group | Control Group | Total
Number analyzed (Participants) | 533 | 528 | 1061
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.5 (8.2) | 59.3 (8.3) | 59.4 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 246 | 257 | 503
  Male | 287 | 271 | 558
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Hong Kong | 468 | 465 | 933
  Malaysia | 65 | 63 | 128

OUTCOME MEASURES:

1. Primary Outcome: Action on Suspected Advanced Liver Fibrosis
Description: Proportion of patients with high fibrosis scores who are referred for specialist care or further liver assessments
Time Frame: Within 1 year of the baseline visit
Population: Patients with abnormal fibrosis scores
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 165 | 131
Participants | 55 | 4

2. Secondary Outcome: Referral for Specialist Care
Description: The proportion of patients referred for specialist care or further liver assessments, regardless of fibrosis score results
Time Frame: Within 1 year of the baseline visit
Population: All participants
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 533 | 528
Participants | 57 | 6

3. Secondary Outcome: Inappropriate Referral for Specialist Care
Description: The proportion of patients with low fibrosis scores who are referred for specialist care. Because NAFLD is highly prevalent and only a minority of patients have advanced fibrosis, referral of patients who will unlikely develop liver-related complications to specialists represents inefficient use of precious healthcare resource and should be minimized. This notion has major resource implications, and the current study will provide important information to guide healthcare policy. We recognize that physicians may have other reasons to refer patients for specialist care (e.g. newly diagnosed viral hepatitis). The reasons for referral will be recorded and reported.
Time Frame: Within 1 year of the baseline visit
Population: Patients with normal fibrosis scores
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 368 | 397
Participants | 1 | 2

4. Secondary Outcome: Confirmed Diagnosis of Advanced Liver Fibrosis
Description: The proportion of patients confirmed to have advanced fibrosis. In this study, a patient is considered to have confirmed advanced fibrosis if (1) liver stiffness measurement by transient elastography is >15 kPa, (2) a liver biopsy shows bridging fibrosis (F3) or cirrhosis (F4), (3) unequivocal radiological features of cirrhosis (cirrhosis with nodular appearance, splenomegaly, ascites or varices), or (4) clinical, radiological or endoscopic evidence of portal hypertension. In case of discrepant results, liver biopsy and unequivocal evidence of cirrhosis and/or portal hypertension will override the liver stiffness measurement results.
Time Frame: Within 1 year of the baseline visit
Population: All participants
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 533 | 528
Participants | 11 | 1

ADVERSE EVENTS:
Time Frame: 1 year
Description: Standard definitions were followed
Arm/Group | Intervention Group | Control Group
All-Cause Mortality (participants affected / at risk) | 9/533 | 3/528
Serious Adverse Events (participants affected / at risk) | 0/533 | 0/528
Other Adverse Events (participants affected / at risk) | 0/533 | 0/528

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-03-27): https://cdn.clinicaltrials.gov/large-docs/75/NCT04241575/Prot_SAP_000.pdf